CLINICAL TRIAL: NCT01359605
Title: An Open-Label, Single-Dose, Study to Assess the Metabolism and Elimination of Varespladib After Oral Administration of [14C]-Labeled Varespladib Methyl in Healthy Male Subjects
Brief Title: Study to Assess the Metabolism and Elimination of [14C]-Labeled Varespladib Methyl in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AN-CVD2215
Record Dates: First submitted 2011-05-19; First posted 2011-05-25 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Healthy Volunteers
Keywords: ADME; Healthy volunteers
MeSH Terms: interventions — varespladib methyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- varespladib methyl (Experimental)
  Interventions: Drug: varespladib methyl

INTERVENTIONS:
Drug: varespladib methyl — 500 mg oral suspension

SUMMARY:
The purpose of the study is to characterize the metabolism and excretion (ADME) of a single oral dose of [14C]varespladib methyl.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent prior to any study specific procedure
* Healthy males, 19 to 55 years of age
* Have a body mass index (BMI) between 18 and 35 kg/m2 inclusive

Exclusion Criteria:

* History or presence of any clinically significant disease or disorder in the opinion of the investigator
* Any clinically relevant abnormal findings in physical examination, clinical chemistry, haematology, urinalysis, or vital signs at baseline in the opinion of the investigator

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Changes in the varespladib blood levels and radioactivity in blood, urine and fecal samples | 1 hour prior to drug, and post dose: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, and 120 hours after drug

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States